CLINICAL TRIAL: NCT01435031
Title: Evaluation of the XIENCE PRIME™ LL and XIENCE Nano™ Everolimus Eluting Coronary Stent Coronary Stents, Performance, and Technique in Chronic Total Occlusions
Brief Title: EXPERT CTO: Evaluation of the XIENCE PRIME™ LL and XIENCE Nano™ Everolimus Eluting Coronary Stent Coronary Stents, Performance, and Technique in Chronic Total Occlusions
Acronym: EXPERT CTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-394
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease (CAD); Chronic Total Occlusion (CTO)
Keywords: Angioplasty; Chronic Total Occlusion (CTO); Chronic total coronary occlusions; Coronary Artery Disease (CAD); Coronary artery stenosis; Total coronary occlusion
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTO Treatment (Other): Subjects receiving at least 1 of the following for the treatment of CTO:
  * XIENCE V® and/or XIENCE nano™ and/or XIENCE PRIME™ LL Everolimus Eluting Coronary Stent
  * HT PROGRESS and/or HT PILOT guide wires in recanalization
  * MINI-TREK Coronary Dilatation Catheter in predilatation
  Interventions: Device: CTO Treatment Device

INTERVENTIONS:
Device: CTO Treatment Device — Subjects receiving at least 1 of the following for the treatment of CTO:
  * XIENCE V® and/or XIENCE nano™ and/or XIENCE PRIME™ LL Everolimus Eluting Coronary Stent
  * HT PROGRESS and/or HT PILOT guide wires in recanalization
  * MINI-TREK Coronary Dilatation Catheter in predilatation

SUMMARY:
A prospective, multi-center, single-arm study to establish the safety and effectiveness of the XIENCE V® Everolimus Eluting Coronary Stent, XIENCE nano™ Everolimus Eluting Coronary Stent, XIENCE PRIME™ LL Everolimus Eluting Coronary Stent, HT PROGRESS and HT PILOT Coronary Guide Wires, and MINI-TREK Coronary Dilatation Catheter in patients undergoing elective percutaneous revascularization of native chronic total coronary occlusions

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is ≥ 18 years of age at the time of consent.
2. Subject is experiencing clinical symptoms considered suggestive of ischemic heart disease (e.g., chest pain or discomfort, heart failure, etc.) or has evidence of myocardial ischemia (e.g., abnormal functional study) attributed to the CTO target vessel and is scheduled for clinically indicated percutaneous revascularization.
3. Subject is eligible and consents to undergo percutaneous coronary intervention (PCI procedure).
4. Subject is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA), stenting, and emergency coronary artery bypass grafting (CABG).
5. Subject is willing and able to sign an informed consent form (ICF) approved by a local Institutional Review Board/Ethics Committee and to follow the protocol with up to 5-year follow up.
6. Female subjects of child-bearing potential must have a negative qualitative or quantitative pregnancy test within 7 days before enrollment and effective birth control must be used up to 1 year following the index procedure.

Angiographic Inclusion Criteria

1. A maximum of one de novo lesion with at least one target segment in a native coronary vessel meeting definition of chronic total occlusion. A "chronic total occlusion" is any non-acute total coronary occlusion fulfilling the following angiographic characteristics and estimated in duration at least 3 months by clinical history and/or comparison with antecedent angiogram or electrocardiogram:

   * High-grade native coronary stenosis
   * TIMI 0 or 1 antegrade flow
2. Occluded segment suitable for placement of coronary stents:

   * Segment without severe tortuosity (angulation ≥ 45º)
   * Segment not located in an excessively distal location

General Exclusion Criteria

Candidates will be excluded from the study if any of the following conditions are present:

1. Patients with any history of allergy to iodinated contrast that cannot be effectively managed medically, or any known allergy to clopidogrel bisulfate (Plavix®), aspirin, heparin, stainless steel, or everolimus
2. Evidence of acute myocardial infarction (MI) within 72 hours of the intended treatment (defined as: Q-wave or non-Q-wave MI having creatine kinase (CK) enzymes 2 × the upper limit of normal (ULN) with the presence of a creatine kinase myocardial-band isoenzyme (CK-MB) above the Institution's ULN, or troponin (I or T) above the Institution's ULN)
3. Previous coronary interventional procedure of any kind within the 30 days prior to the procedure in the target vessel
4. Planned interventional treatment of either the target or any non-target vessel within 30 days post-procedure
5. Planned interventional treatment of either the target or any non-target vessel within 6 months post-procedure with any alternative drug eluting stent (DES) (e.g., CYPHER Sirolimus-Eluting stent, TAXUS Paclitaxel-Eluting stent or Endeavor Zotarolimus-Eluting Endeavor stent)
6. Any contraindication to cardiac catheterization or to any of the standard concomitant therapies used during routine cardiac catheterization and PCI (e.g., aspirin, clopidogrel, unfractionated heparin)
7. Target lesion requires treatment with a device after successful crossing other than PTCA prior to stent placement (including, but not limited to directional or rotational coronary atherectomy, excimer laser, thrombectomy, etc.). Note: Use of alternative technologies to conventional guide wires that are approved by the United States Food and Drug Administration for CTO revascularization (e.g., Asahi Tornus and Corsair catheters, IntraLuminal Therapeutics Safe Cross guide wire, Flowcardia CROSSER system) is permitted and will be collected in the case report form.
8. Patients with history of clinically significant abnormal laboratory findings including:

   * Neutropenia (<1000 neutrophils/mm3) within the previous 2 weeks, or
   * Thrombocytopenia (<100,000 platelets/mm3), or
   * Aspartate Transaminase (AST), Alanine Aminotransferase (ALT), alkaline phosphatase, or bilirubin > 1.5 × ULN, or
   * Serum creatinine > 1.5 mg/dL
9. Patients with evidence of ongoing or active clinical instability including the following:

   * Sustained systolic blood pressure < 100 mmHg or cardiogenic shock
   * Acute pulmonary edema or severe congestive heart failure
   * Suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
   * Suspected dissecting aortic aneurysm
   * Hemodynamically significant valvular heart disease, hypertrophic cardiomyopathy, restrictive cardiomyopathy, or congenital heart disease
10. Target lesion involves a bifurcation including a diseased side branch ≥2.25 mm in diameter that would require treatment
11. Target vessel with a patent bypass graft from prior coronary bypass surgery
12. Proximal coronary stenting of target lesion
13. History of stroke or transient ischemic attack within the prior 6 months
14. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
15. History of bleeding diathesis or coagulopathy or refusal of blood transfusions
16. Patients with any other pathology such as cancer, mental illness, etc., which in the opinion of the Investigator, might put the patient at risk, preclude follow-up, or in any way confound the results of the study.
17. Known previous medical condition yielding expected survival less than 1 year.
18. Patients who are unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements.
19. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; or requires coronary angiography, intravascular ultrasound (IVUS), or other coronary artery imaging procedures

Angiographic Exclusion Criteria

Candidates will be excluded from study if any of the following conditions are met:

1. Occlusion involves segment within previous stent
2. Extensive lesion-related thrombus (TIMI thrombus grade 3 or 4)
3. Previous stenting (drug-eluting or bare metal) in the target vessel unless the following conditions are met:

   * It has been at least 9 months since the previous stenting.
   * That target lesion is at least 15 mm away from the previously placed stent.
   * The previously stented segment (stent plus 5 mm on either side) has no more than 40% diameter stenosis.
4. The target vessel has other lesions proximal to the total occlusion identified with greater than 40% diameter stenosis based on visual estimate or on-line quantitative coronary angiography (QCA). However, planned stenting of the lesion in target vessel which is proximal to the target lesion and can be covered by a single stent (ie, tandem lesions) are acceptable.

Exclusion Criteria (Non-target Lesion):

1. The lesion is located in a native vessel distal to anastomosis with a graft.
2. The vessel has other lesions with greater than 40% diameter stenosis based on visual estimate or on-line QCA.
3. The vessel has evidence of thrombus.
4. The vessel is excessively tortuous.
5. The lesion has any of the following characteristics:

   * Lesion location is aorto-ostial, an unprotected left main lesion, or within 5 mm of the origin of the left anterior descending coronary artery (LAD), left circumflex coronary artery (LCX), or right coronary artery (RCA).
   * Involves a side branch > 2.0 mm in diameter.
   * Is at or distal to a > 45º bend in the vessel.
   * Is moderately to severely calcified.
   * TIMI flow 0 or 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E. Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Kandzari DE, Kini AS, Karmpaliotis D, Moses JW, Tummala PE, Grantham JA, Orr C, Lombardi W, Nicholson WJ, Lembo NJ, Popma JJ, Wang J, Larracas C, Rutledge DR. Safety and Effectiveness of Everolimus-Eluting Stents in Chronic Total Coronary Occlusion Revascularization: Results From the EXPERT CTO Multicenter Trial (Evaluation of the XIENCE Coronary Stent, Performance, and Technique in Chronic Total Occlusions). JACC Cardiovasc Interv. 2015 May;8(6):761-769. doi: 10.1016/j.jcin.2014.12.238. Epub 2015 Apr 22. PMID 25912400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 250 subjects were enrolled in 20 sites from September 13, 2011 to February 7, 2013. Twenty-eight participants were excluded from ITT (N=222) in whom recanalization and pre-dilatation of the target lesion were not completed and/or study stent was not inserted into the coronary guiding catheter.
Pre-assignment Details: ITT set included 222 subjects who met entry criteria, were enrolled in the trial and whose target lesion was successfully crossed and predilated. PP set included all ITT subjects (N = 183) in whom at least 1 study stent was implanted,met procedure success,had follow-up data and had no major protocol deviations due to inappropriate enrollment.
Groups:
- CTO Treatment: Subjects receiving at least 1 of the following for the treatment of CTO:
  * XIENCE V® and/or XIENCE nano™ and/or XIENCE PRIME™ LL Everolimus Eluting Coronary Stent
  * HT PROGRESS and/or HT PILOT guide wires in recanalization
  * MINI-TREK Coronary Dilatation Catheter in predilatation
  CTO Treatment Device: Subjects receiving at least 1 of the following for the treatment of CTO:
  * XIENCE V® and/or XIENCE nano™ and/or XIENCE PRIME™ LL Everolimus Eluting Coronary Stent
  * HT PROGRESS and/or HT PILOT guide wires in recanalization
  * MINI-TREK Coronary Dilatation Catheter in predilatation
Period: ITT at 1 Month
Arm/Group | CTO Treatment
Started | 222 (ITT population)
Completed | 216
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 4
Period: ITT at 6 Months
Arm/Group | CTO Treatment
Started | 216
Completed | 211
Not Completed | 5
Not completed — Death | 2
Not completed — Lost to Follow-up | 3
Period: ITT at 1 Year
Arm/Group | CTO Treatment
Started | 211
Completed | 202
Not Completed | 9
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 6
Period: ITT at 2 Years
Arm/Group | CTO Treatment
Started | 202
Completed | 189
Not Completed | 13
Not completed — Death | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 4
Period: ITT at 3 Years
Arm/Group | CTO Treatment
Started | 189
Completed | 178
Not Completed | 11
Not completed — Death | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 4
Period: ITT at 4 Years
Arm/Group | CTO Treatment
Started | 178
Completed | 171
Not Completed | 7
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: ITT subjects (N=222) include all subjects who met the study entry criteria, signed the written informed consent, were enrolled in the trial and whose target lesion was successfully crossed and predilated.
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.65 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 180
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 178
  More than one race | 17
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 222
Clinical Characteristics [Number; unit: participants]
  Prior Myocardial Infarction (MI) | 61
  Previous Percutaneous Intervention (PCI) | 96
  Prior Coronary Artery Bypass Graft Surgery | 22
  Transient Ischemic Attack (TIA) | 3
  Stroke | 2
  Congestive Heart Failure | 27
  Diabetes Mellitus | 89
  Hypertension | 203
  Dyslipidemia | 215
  Renal Insufficiency/failure | 1
  Atrial fibrillation | 14
  History of bleeding | 18
  Cancer | 4
  Mental Illness | 5
Tobacco use [Number; unit: participants] — Evaluated in 208 subjects.
  participants
    Never used tobacco | 65
    Former user, quit more than 1 month ago | 89
    Current or former, quit within the past month | 54
Number of diseased vessels [Number; unit: participants]
  Single | 170
  Double | 38
  Triple | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stent-related: Major Adverse Cardiac Events (MACE) (Per ITT Set)
Description: The primary stent-related endpoint is MACE, defined as death, MI, or clinically-driven TLR at 1 year post-procedure among all enrolled patients, for whom recanalization and pre-dilatation of the target lesion are completed and the study stent(s) (XIENCE V and/or XIENCE PRIME) is inserted into the coronary guiding catheter.
Time Frame: 1 year
Population: Intention-to-treat (ITT) definition: ITT subjects include all subjects who met the study entry criteria, signed the written informed consent, were enrolled in the trial and whose target lesion was successfully crossed and predilated.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 211
Participants | 39

2. Primary Outcome: Number of Participants With Stent-related: Major Adverse Cardiac Events (MACE) (Per Protocol Set)
Description: as for outcome 1
Time Frame: 1 year
Population: Per-protocol (PP) definition: The per-protocol population is defined as all ITT subjects in whom at least 1 study stent was implanted, met procedure success, had available follow up data (i.e. a MACE event within 360 days or follow up of at least 330 days), and did not have major protocol deviations due to inappropriate enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 183
Participants | 15

3. Primary Outcome: Percentage of Participants With Guide Wire-related: Successful Recanalization of the Chronic Total Occlusion (CTO) (MACE Includes Per ARC Definition of MI)
Description: Successful recanalization of the CTO defined as:
  1. Confirmation of placement of the guide wire in the distal true lumen (component 1)
  2. Absence of in-hospital MACE, based on ARC MI (component 2)
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: All the subjects who met the study entry criteria, signed the written informed consent, were enrolled in the trial and in whom an attempt was made to cross the target lesion with the HT Progress or the HT Pilot guide wires, are included in the ITT population for the guide wire-related analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 138
percentage of participants
  Guide Wire-related Endpoint | 79.0 [71.2 to 85.5]
  Component 1 | 89.9 [83.6 to 94.3]
  Component 2 | 89.1 [82.7 to 93.8]

4. Primary Outcome: Percentage of Participants With Guide Wire-related: Successful Recanalization of the CTO (MACE Includes Per Protocol Definition of MI)
Description: Successful recanalization of the CTO defined as:
  1. Confirmation of placement of the guide wire in the distal true lumen (component 1)
  2. Absence of in-hospital MACE, based on protocol MI (component 2)
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 138
percentage of participants
  Guide Wire-related Endpoint | 87.7 [81 to 92.7]
  Component 1 | 89.9 [83.6 to 94.3]
  Component 2 | 97.8 [93.8 to 99.5]

5. Primary Outcome: Percentage of Participants With Angioplasty Predilatation-related: Successful Predilatation of the CTO
Description: 1. Successful delivery of the MINI-TREK Coronary Dilatation Catheter to and across the target lesion and;
  2. Successful inflation and deflation of the MINI-TREK Coronary Dilatation Catheter and;
  3. Absence of clinically significant vessel perforation, flow-limiting vessel dissection, reduction in thrombolysis in myocardial infarction (TIMI) from baseline or clinically significant arrhythmias requiring medical treatment or device intervention following dilatation with MINI-TREK and;
  4. Achievement of final TIMI flow 3 for the target lesion at the conclusion of the index procedure
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: Angiographically Evaluable Subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 65
percentage of participants | 93.8 [85 to 98.3]

6. Secondary Outcome: Minimum Lumen Diameter (MLD): Pre-procedure
Description: Pre- and post predilatation with the MINI-TREK Coronary Dilatation Catheter.
  MLD is the average of 2 orthogonal views (when possible) of the narrowest point within the area of assessment - in lesion, in stent, or in segment. MLD is visually estimated during angiography by the Investigator; it is measured during Quantitative coronary angiography (QCA) by the Angiographic Core Laboratory.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
mm | 0.01 (0.05)

7. Secondary Outcome: Minimum Lumen Diameter (MLD): Post-procedure
Description: Pre- and post predilatation with the MINI-TREK Coronary Dilatation Catheter.
  MLD is the average of 2 orthogonal views (when possible) of the narrowest point within the area of assessment - in lesion, in stent, or in segment. MLD is visually estimated during angiography by the Investigator; it is measured during QCA by the Angiographic Core Laboratory.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CTO Treatment
Number analyzed (Participants) | 221
mm
  In-Segment | 1.85 (0.47)
  In-Stent | 2.32 (0.39)

8. Secondary Outcome: Percentage of Participants With Change in Thrombolysis in Myocardial Infarction (TIMI) Flow Grade: Pre-procedure
Description: Pre- and post predilatation with the MINI-TREK Coronary Dilatation Catheter.
  TIMI Classification:
  TIMI 0 No perfusion.
  TIMI 1 Penetration with minimal perfusion. Contrast fails to opacify the entire bed distal to the stenosis for the duration of the cine run.
  TIMI 2 Partial perfusion. Contrast opacifies the entire coronary bed distal to the stenosis. However, the rate of entry and/or clearance is slower in the coronary bed distal to the obstruction than in comparable areas not perfused by the dilated vessel.
  TIMI 3 Complete perfusion. Filling and clearance of contrast equally rapid in the coronary bed distal to stenosis as in other coronary beds.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set.The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
percentage of participants
  0 | 95.9 [92.4 to 98.1]
  1 | 3.6 [1.6 to 7.0]
  2 | 0.0 [0.0 to 1.6]
  3 | 0.5 [0.0 to 2.5]

9. Secondary Outcome: Percentage of Participants With Change in TIMI Flow Grade: Post-procedure
Description: as for outcome 8
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 221
percentage of participants
  0 | 0.5 [0.0 to 2.5]
  1 | 0.0 [0.0 to 1.7]
  2 | 1.8 [0.5 to 4.6]
  3 | 97.7 [94.8 to 99.3]

10. Secondary Outcome: Percentage of Participants With Device Success
Description: Achievement of <50% diameter stenosis within the target lesion segment using assigned study device
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 221
percentage of participants | 100 [98.3 to 100]

11. Secondary Outcome: Percentage of Participants With Procedure Success
Description: Device success and absence of in-hospital MACE.
  Per-protocol MI definition: Myocardial infarctions per protocol definition were categorized as Q-wave (development of new, pathological Q waves on the ECG) or non-Q-wave (elevation of CK levels to greater than two times the upper limit of normal and elevated CK-MB in the absence of new pathological Q waves).
  Per ARC MI definition: Myocardial infarctions per ARC definition were also categorized as Q-wave (development of new pathological Q waves in 2 or more contiguous leads (according to the Minnesota code) with or without post-procedure CK or CK-MB levels elevated above normal) or non-Q-wave (all MIs not classified as Q-wave). ARC defined MIs were further classified as Periprocedural PCI, Periprocedural CABG, Spontaneous, Sudden Death, and Reinfarction based on biomarker and additional criteria and as ST Elevation MI (STEMI) or Non-ST Elevation MI (NSTEMI) based on ST segment.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 221
percentage of participants
  Per Protocol MI definition | 96.4 [93.0 to 98.4]
  Per ARC MI definition | 89.6 [84.8 to 93.3]

12. Secondary Outcome: Percentage of Participants With Procedural Success With Antegrade Crossing
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set. The number of participants analyzed include the numbers of subjects with corresponding crossing method that were evaluable for procedural success.
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 187
percentage of participants | 97.9

13. Secondary Outcome: Percentage of Participants With Procedural Success With Subintimal Tracking and Re-entry (STAR) Technique
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 7
percentage of participants | 100

14. Secondary Outcome: Percentage of Participants With Procedural Success With Knuckle Wire
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 1
percentage of participants | 100.0

15. Secondary Outcome: Percentage of Participants With Procedural Success With Primary Retrograde Wire Crossing
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 12
percentage of participants | 91.7

16. Secondary Outcome: Percentage of Participants With Procedural Success With Controlled Antegrade-Retrograde Technique (CART)
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 1
percentage of participants | 100

17. Secondary Outcome: Percentage of Participants With Procedural Success With Reverse CART
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 9
percentage of participants | 77.8

18. Secondary Outcome: Percentage of Participants With Procedural Success With Kissing Wire Technique
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set.The number of participants analyzed include the numbers of subjects with corresponding crossing method that were evaluable for procedural success.
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 1
percentage of participants | 100

19. Secondary Outcome: Percentage of Participants With Procedural Success With Sub Intimal Technique
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique.
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 1
percentage of participants | 100.0

20. Secondary Outcome: Percentage of Participants With Procedural Success With Multiple Crossing Techniques
Description: Defined as device success and absence of in-hospital MACE with antegrade crossing technique
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 5
percentage of participants | 80.0

21. Secondary Outcome: Resource Utilization: Procedural Time
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Minutes | 79.88 (48.5)

22. Secondary Outcome: Resource Utilization: Fluoroscopic Time
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Minutes | 33.61 (23.29)

23. Secondary Outcome: Resource Utilization: Contrast Volume
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT set.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
mL | 259.00 (136.74)

24. Secondary Outcome: Percentage of Participants With Clinically Significant Perforation
Description: Any perforation resulting in hemodynamic instability and/or requiring intervention including pericardiocentesis, embolization, prolonged balloon occlusion, stent graft or comparable therapy
Time Frame: Participants were monitored for the duration of index procedure, an average of 79.9 ± 48.5 minutes
Population: ITT Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
percentage of participants
  Post Last Mini-Trek Balloon Angiography (n=67) | 0.0 [0.0 to 5.4]
  Final Angiography (n=221) | 0 [0.0 to 1.7]
  Site reported (n=222) | 0.0 [0.0 to 1.6]

25. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 219
Participants | 8

26. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 215
Participants | 13

27. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 211
Participants | 21

28. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
  The overall number of participants analysed include ITT subjects who experienced the specific event within 720 days or ITT subjects with follow-up of at least 690 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 205
Participants | 32

29. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
  The overall number of participants analysed include ITT subjects who experienced the specific event within 1080 days or ITT subjects with follow-up of at least 1050 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 199
Participants | 37

30. Secondary Outcome: Number of Participants With Major Adverse Cardiac Events (MACE)
Description: Per protocol. Defined as death, MI (Q wave and non-Q wave) or clinically-driven target lesion revascularization.
Time Frame: 4 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
  The overall number of participants analysed include ITT subjects who experienced the specific event within 1440 days or ITT subjects with follow-up of at least 1410 days.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 196
Participants | 44

31. Secondary Outcome: Number of Participants Experiencing Death
Description: MACE Component; per protocol.
  Death is divided into 2 categories:
  Cardiac death is defined as death due to any of the following:
  1. Acute MI
  2. Cardiac perforation/pericardial tamponade
  3. Arrhythmia or conduction abnormality
  4. Stroke within 30 days of the procedure or stroke suspected of being related to the procedure
  5. Death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery
  6. Any death in which a cardiac cause cannot be excluded.
  Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 1

32. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 31
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 214
Participants | 3

33. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 31
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 210
Participants | 4

34. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 31
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 202
Participants | 11

35. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 31
Time Frame: 3 years
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 195
Participants | 16

36. Secondary Outcome: Number of Participants Experiencing Death
Description: as for outcome 31
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 191
Participants | 20

37. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: TLF component.
  Cardiac death was defined as death due to any of the following:
  1. Acute MI
  2. Cardiac perforation/pericardial tamponade
  3. Arrhythmia or conduction abnormality
  4. Stroke within 30 days of the procedure or stroke suspected of being related to the procedure
  5. Death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery
  6. Any death in which a cardiac cause cannot be excluded
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 1

38. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: as for outcome 37
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 212
Participants | 1

39. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: as for outcome 37
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 208
Participants | 2

40. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: as for outcome 37
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 196
Participants | 5

41. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: as for outcome 37
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 188
Participants | 8

42. Secondary Outcome: Number of Participants Experiencing Cardiac Death
Description: as for outcome 37
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 181
Participants | 10

43. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: MACE Component;
  Myocardial Infarction (per ARC definition)
  * Q wave MI: Development of new pathological Q waves in 2 or more contiguous leads with or without post-procedure CK or CK-MB levels elevated above normal
  * Non-Q-wave MI: All MIs not classified as Q-wave.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 219
Participants | 24

44. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: as for outcome 43
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 213
Participants | 26

45. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: as for outcome 43
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 209
Participants | 29

46. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: as for outcome 43
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 197
Participants | 31

47. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: as for outcome 43
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 188
Participants | 34

48. Secondary Outcome: Number of Participants With Myocardial Infarction Q Wave and Non-Q Wave (MI)
Description: as for outcome 43
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 182
Participants | 37

49. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: TLF Component; per ARC
  Target vessel-related MI: All infarcts that cannot be clearly attributed to a vessel other than the target vessel will be considered related to the target vessel.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 219
Participants | 23

50. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: as for outcome 49
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 213
Participants | 24

51. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: as for outcome 49
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 209
Participants | 25

52. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: as for outcome 49
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 197
Participants | 27

53. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: as for outcome 49
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 188
Participants | 28

54. Secondary Outcome: Number of Participants With Target Vessel-related MI
Description: as for outcome 49
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 181
Participants | 28

55. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat percutaneous coronary intervention (PCI) or Coronary artery bypass graft (CABG) to the target lesion/site.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 2

56. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat PCI or CABG to the target lesion/site.
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 212
Participants | 5

57. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat PCI or CABG to the target lesion/site.
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 207
Participants | 13

58. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat PCI or CABG to the target lesion/site.
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 194
Participants | 18

59. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat PCI or CABG to the target lesion/site.
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 185
Participants | 19

60. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Repeat PCI or CABG to the target lesion/site.
Time Frame: 4 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 177
Participants | 21

61. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: TLF and MACE component. Revascularization at the target lesion associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis >= 50% by QCA, or revascularization of a target lesion with diameter stenosis >= 70% by QCA without either angina or a positive functional study.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 2

62. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: as for outcome 61
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 212
Participants | 5

63. Secondary Outcome: Number of Participants With Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: as for outcome 61
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 207
Participants | 13

64. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: as for outcome 61
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 194
Participants | 18

65. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: as for outcome 61
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 185
Participants | 19

66. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (Clinically-Driven TLR)
Description: as for outcome 61
Time Frame: 4 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 177
Participants | 20

67. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: Repeat PCI or CABG of the target vessel. Revascularization in the target vessel associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis >= 50% by QCA, or revascularization of a target vessel with diameter stenosis >= 70% by QCA without either angina or a positive functional study
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 2

68. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 67
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 212
Participants | 6

69. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 67
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 207
Participants | 15

70. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 67
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 194
Participants | 21

71. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 67
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 185
Participants | 22

72. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 67
Time Frame: 4 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 177
Participants | 24

73. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Composite endpoint comprised of cardiac death, target vessel MI, or clinically-driven target vessel revascularization. Per protocol.
  Target vessel failure will be reported when any of the following events occur:
  * Recurrent MI occurs in territory not clearly attributed to a vessel other than the target vessel.
  * Cardiac death not clearly due to a non-target vessel endpoint.
  * Target vessel revascularization is determined.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 219
Participants | 8

74. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 73
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 213
Participants | 12

75. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 73
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 209
Participants | 21

76. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 73
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 199
Participants | 29

77. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 73
Time Frame: 3 years
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 192
Participants | 32

78. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 73
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 186
Participants | 36

79. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR. Per protocol.
Time Frame: 30 days
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 219
Participants | 8

80. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR. Per protocol.
Time Frame: 6 months
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 213
Participants | 11

81. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR. Per protocol.
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 209
Participants | 19

82. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 199
Participants | 26

83. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR
Time Frame: 3 years
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 192
Participants | 29

84. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: Composite of cardiac death, target vessel-related MI, and clinically-driven TLR
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 186
Participants | 32

85. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Academic Research Consortium (ARC) criteria; definite and probable
  Definite stent thrombosis as defined by ARC criteria: Angiographic confirmation with at least one of the following: Acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy).
  Probable stent thrombosis as defined by ARC criteria: Any unexplained death within the first 30 days or, regardless of the time after the index procedure, any MI related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause.
Time Frame: Acute (0-24 hours)
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Participants | 0

86. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Academic Research Consortium (ARC) criteria; definite and probable. Definite stent thrombosis as defined by ARC criteria: Angiographic confirmation with at least one of the following: Acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy).
  Probable stent thrombosis as defined by ARC criteria: Any unexplained death within the first 30 days or, regardless of the time after the index procedure, any MI related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause.
Time Frame: Subacute (>24 hours to 30 days)
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 218
Participants | 2

87. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: as for outcome 86
Time Frame: Late (>30 days to 1 year)
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 206
Participants | 1

88. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: as for outcome 86
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 207
Participants | 3

89. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Academic Research Consortium (ARC) criteria.
  Definite stent thrombosis as defined by ARC criteria: angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic ECG changes that suggest acute ischemia or typical rise and fall of cardiac biomarkers OR pathological confirmation at autopsy or via examination of tissue retrieved following thrombectomy).
  Probable stent thrombosis as defined by ARC criteria: any unexplained death within the first 30 days or, regardless of the time after the index procedure, any MI related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation and in the absence of any other obvious cause.
Time Frame: 2 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 192
Participants | 3

90. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: as for outcome 89
Time Frame: 3 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 182
Participants | 3

91. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: as for outcome 89
Time Frame: 4 years
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 174
Participants | 3

92. Secondary Outcome: Number of Participants With Occurrence of Stent Fracture at Target Lesion
Description: Assessed by fluoroscopy in patients undergoing clinically-driven angiographic follow-up.
Time Frame: 1 year
Population: ITT set. The number of participants analyzed include subjects who had available follow up data at that time frame.
  The overall number of participants analysed include ITT subjects who experienced the specific event within 360 days or ITT subjects with follow-up of at least 330 days
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Participants | 0.0

93. Secondary Outcome: Number of Participants With Occurrence of Stent Fracture at Target Lesion
Description: Assessed by fluoroscopy in patients undergoing clinically-driven angiographic follow-up.
Time Frame: 2 years
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Participants | 0.0

94. Secondary Outcome: Number of Participants With Occurrence of Stent Fracture at Target Lesion
Description: Assessed by fluoroscopy in patients undergoing clinically-driven angiographic follow-up.
Time Frame: 3 years
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Participants | 0.0

95. Secondary Outcome: Number of Participants With Occurrence of Stent Fracture at Target Lesion
Description: Assessed by fluoroscopy in patients undergoing clinically-driven angiographic follow-up.
Time Frame: 4 years
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | CTO Treatment
Number analyzed (Participants) | 222
Participants | 0.0

ADVERSE EVENTS:
Time Frame: 4 years
Description: ITT set
Arm/Group | CTO Treatment
All-Cause Mortality (participants affected / at risk) | 20/222
Serious Adverse Events (participants affected / at risk) | 92/222
Other Adverse Events (participants affected / at risk) | 141/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTO Treatment (N=222)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 20
Angina unstable (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 6
Coronary artery dissection (Cardiac disorders) | 6
Coronary artery occlusion (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 2
Coronary artery thrombosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 5
Myocardial ischaemia (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 4
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Catheter site haematoma (General disorders) | 1
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 4
Device malfunction (General disorders) | 1
Fatigue (General disorders) | 1
Medical device complication (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Thrombosis in device (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Chest wall abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 3
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Cardiac enzymes increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Haemorrhage intracranial (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Nephropathy (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic dissection (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Intermittent claudication (Vascular disorders) | 2
Ischaemia (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTO Treatment (N=222)
Anaemia (Blood and lymphatic system disorders) | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 8
Angina pectoris (Cardiac disorders) | 32
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 7
Atrial flutter (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 5
Coronary artery dissection (Cardiac disorders) | 18
Coronary artery perforation (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 3
Ventricular tachycardia (Cardiac disorders) | 7
Cushing's syndrome (Endocrine disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Mesenteric artery stenosis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Catheter site haematoma (General disorders) | 13
Catheter site haemorrhage (General disorders) | 1
Catheter site pain (General disorders) | 7
Catheter site related reaction (General disorders) | 1
Chest pain (General disorders) | 2
Fatigue (General disorders) | 4
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site haemorrhage (General disorders) | 1
Non-cardiac chest pain (General disorders) | 13
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Thrombosis in device (General disorders) | 2
Bile duct stenosis (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Wound infection (Infections and infestations) | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 5
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Blood creatine phosphokinase MB increased (Investigations) | 2
Cardiac enzymes increased (Investigations) | 5
Cardiac stress test abnormal (Investigations) | 1
Electrocardiogram QRS complex abnormal (Investigations) | 1
Oxygen consumption decreased (Investigations) | 1
Smear cervix abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Lactic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 5
Renal failure (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 10
Intermittent claudication (Vascular disorders) | 5
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1
Angina unstable (Cardiac disorders) | 5
Atrioventricular block second degree (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 6
Coronary artery occlusion (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 2
Coronary artery thrombosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 5
Pulseless electrical activity (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Device malfunction (General disorders) | 1
Medical device complication (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chest wall abscess (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Haemorrhage intracranial (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Nephropathy (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic dissection (Vascular disorders) | 2
Arteriosclerosis (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days